CLINICAL TRIAL: NCT05576259
Title: oVRcome - Self Guided Virtual Reality for Social Anxiety Disorder. A Randomised Controlled Trial.
Brief Title: oVRcome - Self Guided Virtual Reality for Social Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Otago (Other)
Collaborators: oVRcome (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: oVRcome social anxiety 1.2
Record Dates: First submitted 2022-10-09; First posted 2022-10-12 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2023-11

CONDITIONS: Social Anxiety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Smartphone application (app) in combination with headset (Experimental): The intervention oVRcome is self-help VRET for social anxiety, that is delivered through a smartphone application (app) in combination with headset that holds the smartphone and uses 360º video. oVRcome includes 6 modules of psychoeducation, relaxation, mindfulness, cognitive techniques, exposure through VR, and a relapse prevention module which are aimed to be completed weekly.
  Interventions: Other: oVRcome phone app with headset
- Waitlist (No Intervention): Participants in the waitlist condition will be offered the intervention directly after post-test.

INTERVENTIONS:
Other: oVRcome phone app with headset — The intervention oVRcome is self-help VRET for social anxiety, that is delivered through a smartphone application (app) in combination with headset that holds the smartphone and uses 360º video. oVRcome includes 6 modules of psychoeducation, relaxation, mindfulness, cognitive techniques, exposure through VR, and a relapse prevention module which are aimed to be completed weekly.
  Arms: Smartphone application (app) in combination with headset

SUMMARY:
Social anxiety is characterised by excessive fear of being negatively judged, embarrassed or humiliated during social interactions and is common with a lifetime prevalence of 12.1%. Cognitive behavioural therapy is the first line of treatment, but people may not seek treatment due to a number of factors including the discomfort experienced in seeking help, inconvenience, and the experience of psychotherapy itself. With Virtual Reality (VR), users can have increased control in how gradually they expose themselves to social situations. In studies of VR in people with specific phobias, 76% of people prefer VR exposure to in vivo exposure. There is emerging evidence for the use of VR in social phobia.

oVRcome, is a self-help VRET for social anxiety symptoms and specific phobias, that is delivered through a smartphone application (app) in combination with a low cost headset that holds the smartphone and uses 360º video.

This study will evaluate the effectiveness of the oVRcome social anxiety program for social anxiety symptoms. We hypothesize that oVRcome will reduce social anxiety symptom severity over a 6-week treatment period compared to waiting-list control

ELIGIBILITY:
Inclusion Criteria:

* are between 18-64 years old
* have moderate (or higher) social anxiety disorder symptoms on Liebowitz social anxiety scale (>60)
* have access to a smart phone and internet
* willing to participate in the research study and providing informed consent

Exclusion Criteria:

* present with symptoms of severe depression or suicidality respectively as measured with the PHQ-9; total score > 19, =3 on suicidality item
* have insufficient knowledge of the English language
* are under current treatment for social phobia or psychotropic medication (unless on stable dosage for the previous 3 months and no changes planned during the study period).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-10-08 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Liebowitz social anxiety scale -self report (LSAS) | Week 6
  Assesses the way that social phobia plays a role in participants life across a variety of situations. Higher scores indicate more severe symptoms. Min 0 Max 144

SECONDARY OUTCOMES:
Brief Fear of Negative Evaluation Scale | week 0,6,12,18
  Scores range from 1 through to 60 with higher scores indicating higher fear of negative evaluation
Patient's Global Impressions of Improvement (PGI-I) scale | Week 1,2,3,4,5,6,7,8,9,10,11,12,18
  Assesses patients' overall perception of their condition in a 1-item questionnaires that ask an individual patient to rate the perceived change in his/her condition in response to therapy at endpoint. Min 1 (very much improved) Max 7 (very much worse).
Patient Health Questionnaire - PHQ 9 | Week 0,6,12,18
  PHQ-9 scores range from 0 through to 27, with higher scores indicating more severe depressive symptoms
Modified Gatineau Presence Questionnaire First item | Week 4,5,6
  Assess degree of realism using virtual reality. Scores range from 1 (very realistic) through to 100 (not very realistic)
Fast Motion Sickness Scale (FMS) | Week 4,5,6
  Measures motion sickness with virtual reality. Scores range from zero (no sickness at all) to 20 (frank sickness).
Changes in behaviour that may have been previously avoided because of the phobia | Week 6,12,18
  Free text response

CONTACTS AND LOCATIONS:
Overall Officials: Cameron Lacey, PhD, Principal Investigator — University of Otago, Christchurch
Locations (1):
- University of Otago, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lacey C, Frampton C, Beaglehole B. A self-guided virtual reality solution for social anxiety: Results from a randomized controlled study. J Psychiatr Res. 2024 Dec;180:333-339. doi: 10.1016/j.jpsychires.2024.10.032. Epub 2024 Nov 4. PMID 39515186
- See also: Related Info — http://ovrcome.io